

FOR IRB USE ONLY IRB ID #: 202004074 APPROVAL DATE: 04/05/21 RELEASED DATE: 04/05/21 EXPIRATION DATE: 04/04/22

## VERBAL ASSENT INFORMATION SHEET

Project Title: **Piloting Virtual Reality** 

Investigator(s): Ellen Fitzsimmons-Craft, PHD

We are doing a research study. A research study is a special way to find out about something. We are trying to compare different digital technologies that teach about healthy habits to see which one is more helpful for kids.

If you decide that you want to be in this study, this is what will happen. You and your parents will come into our office to try one of the educational digital technologies we're testing. We will ask you some questions before and after you try the technology to see how you liked it and how it affected you. We will send you and your parents some questions to answer two weeks later to see how the technology affected you over those two weeks..

We want to tell you about some things that might hurt or upset you if you are in this study. Using the digital technologies could make you feel sad or upset, but we'll provide your family with resources for seeking help if you need it. If you get assigned to the technology that requires more moving around, you might run into something while you're using it, but someone will be in the room with you to try to keep you from doing that, and we'll make sure there aren't many things around for you to run into. If you get assigned to the technology that requires more moving around it might make you experience motion sickness, like in a car. If this happens you can stop playing.

We don't know if being in this research study will help you. But we hope to learn something that will help other people someday.

When we are done with the study, we will write a report about what we found out. We won't use your name in the report.

You don't have to be in this study. It's up to you. If you say okay now, but you change your mind later, that's okay too. All you have to do is tell us.